CLINICAL TRIAL: NCT01064479
Title: A Randomized, Placebo-Controlled, Phase 2 Study of Docetaxel and Cisplatin/Carboplatin With or Without Erlotinib in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: Combination Chemotherapy With or Without Erlotinib Hydrochloride in Treating Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-0395; NCI-2011-03782 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0395 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Squamous Cell Carcinoma of the Hypopharynx; Metastatic Squamous Cell Carcinoma of the Larynx; Metastatic Squamous Cell Carcinoma of the Oral Cavity; Metastatic Squamous Cell Carcinoma of the Oropharynx; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage IV Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IV Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IV Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IV Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVB Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVC Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (combination chemotherapy and erlotinib hydrochloride) (Experimental): Patients receive docetaxel IV over 1 hour and cisplatin IV over 2 hours or carboplatin IV over 2 hours on day 1 and erlotinib hydrochloride PO daily on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression and unacceptable toxicity. Patients achieving complete response, partial response, or stable disease may continue erlotinib hydrochloride treatment.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Docetaxel; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment
- Arm B (combination chemotherapy and placebo) (Active Comparator): Patients receive docetaxel and cisplatin or carboplatin as in Arm I and placebo PO daily on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression and unacceptable toxicity. Patients achieving complete response, partial response, or stable disease may continue placebo treatment.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
  Arms: Arm A (combination chemotherapy and erlotinib hydrochloride)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Pharmacological Study — Optional correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm B (combination chemotherapy and placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase II trial studies how well combination chemotherapy with or without erlotinib hydrochloride works in treating patients with squamous cell carcinoma of the head and neck that has spread to other parts of the body or has come back. Drugs used in chemotherapy, such as docetaxel, cisplatin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy with or without erlotinib hydrochloride may be an effective treatment for squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the efficacy of adding erlotinib hydrochloride (erlotinib) to chemotherapy to improve progression free survival in patients with metastatic or recurrent squamous cell carcinoma of the head and neck.

SECONDARY OBJECTIVES:

I. Evaluate overall survival, response rate, disease control rate, and duration of response by treatment with or without erlotinib.

II. Evaluate quality of life (patient reported outcomes) by treatment with or without erlotinib.

III. Evaluate the safety profile of erlotinib in combination with chemotherapy. IV. Correlate the occurrence of erlotinib-induced rash with outcomes. V. To evaluate the steady-state pharmacokinetics of erlotinib. VI. To explore the prognostic and predictive value of epidermal growth factor receptor related biomarkers and other biomarkers, including blood and tissue proteomic and blood and tissue genomic markers, that may be associated with clinical outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive docetaxel intravenously (IV) over 1 hour and cisplatin IV over 2 hours or carboplatin IV over 2 hours on day 1, and erlotinib hydrochloride orally (PO) daily on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression and unacceptable toxicity. Patients achieving complete response, partial response, or stable disease may continue erlotinib hydrochloride treatment.

ARM B: Patients receive docetaxel and cisplatin or carboplatin as in Arm I and placebo PO daily on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression and unacceptable toxicity. Patients achieving complete response, partial response, or stable disease may continue placebo treatment.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or recurrent squamous cell carcinoma of the head and neck (SCCHN) of the oral cavity, oropharynx, hypopharynx or larynx; metastatic or recurrent lesions of the nasopharynx and sinus are excluded
* Radiologically measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan; measurable lymph nodes are required to be >= 15 mm in size (short axis diameter)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Total bilirubin =< upper limit of normal (ULN) (excluding Gilbert's disease)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Serum creatinine =< 1.5 x ULN
* Patients with reproductive potential (e.g., females menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures for the duration of study drug therapy and for at least 30 days after completion of study drug therapy; female patients of childbearing potential must provide a negative pregnancy test (serum or urine) =< 14 days prior to treatment initiation
* Written informed consent to participate in the study according to the investigational review board (IRB) or independent ethics committee (IEC)

Exclusion Criteria:

* Histology other than squamous cell carcinoma
* Primary sites other than oral cavity, oropharynx, hypopharynx, and larynx
* Prior palliative chemotherapy for metastatic or recurrent disease
* Prior biological therapy for metastatic or recurrent disease within 3 weeks prior to randomization
* Patients with known, untreated brain metastases; patients with treated (irradiated or resected) brain metastases are eligible if treatment was completed more than 28 days prior to study entry and if clinical neurologic function is stable
* Pre-existing peripheral neuropathy >= grade 2
* History of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g., Crohn's disease, ulcerative colitis); patients requiring feeding tubes are permitted
* Other active malignancies requiring chemotherapy treatment within 2 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical or breast cancer or superficial, resected melanoma
* Serious underlying medical condition which would impair the ability of the patient to receive protocol treatment, in the opinion of the treating physician
* History of allergic reactions to compounds of similar chemical composition to the study drugs (docetaxel, cisplatin, carboplatin, erlotinib or their excipients), or other drugs formulated with polysorbate 80
* Any concurrent anti-cancer therapy, excluding hormonal therapy for prostate or breast cancer
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent
* Women who are pregnant or breast-feeding and women or men not practicing effective birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-02-05 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiuning Le, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with histologically confirmed metastatic or recurrent SCCHN of the oral cavity, oropharynx, hypopharynx or larynx who have an ECOG performance status of 0-2, measurable disease and no prior chemotherapy for their metastatic or recurrent disease were enrolled
Pre-assignment Details: 123 participants registered-4 participants were inevaluable (2 refused not due to toxicity, 2 other).
Period: Overall Study
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo)
Started | 60 | 59
Completed | 45 | 42
Not Completed | 15 | 17
Not completed — Death | 10 | 11
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Disease progression | 1 | 1
Not completed — Toxicity | 1 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo) | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 51 | 103
  >=65 years | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 47 | 45 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race and ethnicity were reported for participants. The data collected was for all participants and not separated in each arm.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 4 | 6
    White | 51 | 49 | 100
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Kaplan-Meier methods will be used to summarize PFS. In the primary analysis, differences in PFS in Arm A versus Arm B will be tested using a stratified log-rank test with a two-sided alpha of 0.10. Hazard ratios for PFS will be presented using point estimates and 95% confidence intervals.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo)
Number analyzed (Participants) | 60 | 59
months | 6.08 [5.45 to 7.52] | 4.4 [3.45 to 5.78]

2. Secondary Outcome: Overall Survival (OS)
Description: Kaplan-Meier methods will be used to summarize OS. Hazard ratios for OS will be presented using point estimates and 95% confidence intervals.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo)
Number analyzed (Participants) | 60 | 59
months | 16.95 [10.12 to NA] — below the level of detection | 13.67 [10.64 to 18.73]

3. Secondary Outcome: Number of Participants With Tumor Response (Complete Response [CR] + Partial Response [PR])
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo)
Number analyzed (Participants) | 60 | 59
Participants
  Complete Response | 4 | 5
  Partial Response | 27 | 19
  Progressive Disease | 8 | 13
  Stable Disease | 16 | 17
  Inevaluable | 5 | 5

4. Secondary Outcome: Disease Control (CR + PR + Stable Disease [SD])
Description: Complete Response (CR) + Partial Response (PR) + Stable disease
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo)
Number analyzed (Participants) | 60 | 59
Participants | 47 | 41

5. Secondary Outcome: Rash Rates
Description: Participants with a Rash of at least grade 2 within cycle 1.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo)
Number analyzed (Participants) | 60 | 59
Participants | 20 | 4

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last does of study medication, up to 5 years
Description: MedDRA v12
Arm/Group | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) | Arm B (Combination Chemotherapy and Placebo)
All-Cause Mortality (participants affected / at risk) | 37/60 | 53/59
Serious Adverse Events (participants affected / at risk) | 21/60 | 46/59
Other Adverse Events (participants affected / at risk) | 56/60 | 55/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) (N=60) | Arm B (Combination Chemotherapy and Placebo) (N=59)
Nausea (Gastrointestinal disorders) | 4 | 2
Oral pain (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 1
Syncope (Nervous system disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Dehydration (Gastrointestinal disorders) | 8 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Lung infection (Infections and infestations) | 7 | 5
Skin infection (Infections and infestations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 3
Stroke (Nervous system disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 3 | 0
Fever (General disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Esophageal ulcer (Gastrointestinal disorders) | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Stoma site infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 2
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Catheter related infection (Injury, poisoning and procedural complications) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Asystole (Cardiac disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Oral cavity fistula (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Hyponatremia (Investigations) | 1 | 1
Hypokalemia (Investigations) | 1 | 0
Infections and infestations-other (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Combination Chemotherapy and Erlotinib Hydrochloride) (N=60) | Arm B (Combination Chemotherapy and Placebo) (N=59)
Dehydration (Metabolism and nutrition disorders) | 10 | 4
Diarrhea (Gastrointestinal disorders) | 46 | 30
Anemia (Blood and lymphatic system disorders) | 13 | 4
Nausea (Gastrointestinal disorders) | 38 | 27
Fatigue (General disorders) | 40 | 33
Mucositis oral (Gastrointestinal disorders) | 16 | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 35 | 12
Anorexia (Metabolism and nutrition disorders) | 14 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 22 | 13
Pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Vomiting (Gastrointestinal disorders) | 23 | 10
Rash acneform (Skin and subcutaneous tissue disorders) | 31 | 10
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Oral pain (Gastrointestinal disorders) | 11 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 12
Constipation (Gastrointestinal disorders) | 6 | 11
Dizziness (Nervous system disorders) | 7 | 10
Weight loss (Investigations) | 10 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 9
Nail discoloration (Skin and subcutaneous tissue disorders) | 6 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Hypomagnesemia (Investigations) | 4 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 4
Watering eyes (Eye disorders) | 6 | 2
Blood bilirubin increase (Investigations) | 5 | 0
Blurred vision (Eye disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 6
Dysphagia (Gastrointestinal disorders) | 4 | 3
Edema face (General disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Eyelid function disorder (Eye disorders) | 3 | 1
Fever (General disorders) | 5 | 0
Hypokalemia (Investigations) | 7 | 2
Hyponatriema (Investigations) | 6 | 1
Lung infection (Infections and infestations) | 3 | 2
Mucosal infection (Infections and infestations) | 0 | 4
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 3
Palmar-plantar erythrodysesthesia syndrom (Skin and subcutaneous tissue disorders) | 2 | 3
Paresthesia (Nervous system disorders) | 1 | 3
Paronychia (Infections and infestations) | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2
Platelet count decreased (Investigations) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rash pustular (Skin and subcutaneous tissue disorders) | 3 | 1
Skin infection (Infections and infestations) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT01064479/Prot_SAP_000.pdf